CLINICAL TRIAL: NCT01168492
Title: Analgesia During Pediatric Digestive Endoscopy: a Comparison of Two Protocols for Procedural Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Denise Herzog, Associate Professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: cme#2857
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Pain
Keywords: pediatric; gastroscopy; colonoscopy; sedation; ketamine
MeSH Terms: conditions — Pain | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ketamine (Experimental): group with triple sedation (ketamine, midazolam, meperidine)
  Interventions: Drug: ketamine
- placebo (Placebo Comparator): group with conventional sedation and placebo ( midazolam, meperidine and placebo)
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: ketamine — 0.5mg/kg ketamine iv
  Other Names: no other names

SUMMARY:
The purpose of this study is to determine whether ketamine, midazolam, and meperidine are more effective than midazolam and meperidine alone for procedural sedation and analgesia in pediatric digestive endoscopy. Secondary outcomes are the incidence of cardiorespiratory side effects and the necessity of rescue doses.

DETAILED DESCRIPTION:
90 patients will be included. The sedation will include 0.1mg/kg, max 5mg iv of midazolam, 1mg/kg, max 50mg iv of meperidine, and placebo (0.9%NaCl) or ketamine 0.5mg/kg iv. Rescue doses will be given as usual, using meperidine and or midazolam 50% of the initial dose.

ELIGIBILITY:
Inclusion Criteria:

* Children =/> 10 years of age
* Undergoing elective diagnostic colonoscopy
* ASA score class 1-3.

Exclusion Criteria:

* Children younger than 10 years of age
* Known epilepsy under treatment
* ASA score class 4 or more
* Interventional colonoscopy (e.g.polypectomy)

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2010-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
pain score | after one year
  pain scores are accorded at the end of each endoscopy. Pain scores of the two groups will be compared after one year

SECONDARY OUTCOMES:
necessity of cardiopulmonary intervention (Oxygen requirements) | after one year
  according to Observer'sAssessment of Alertness/Sedation (OAAS) score

CONTACTS AND LOCATIONS:
Overall Officials: Denise Herzog, MD, Principal Investigator — Université de Montréal
Locations (1):
- Sainte Justine Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Gilger MA, Spearman RS, Dietrich CL, Spearman G, Wilsey MJ Jr, Zayat MN. Safety and effectiveness of ketamine as a sedative agent for pediatric GI endoscopy. Gastrointest Endosc. 2004 May;59(6):659-63. doi: 10.1016/s0016-5107(04)00180-4. PMID 15114309
- [Background] McQuaid KR, Laine L. A systematic review and meta-analysis of randomized, controlled trials of moderate sedation for routine endoscopic procedures. Gastrointest Endosc. 2008 May;67(6):910-23. doi: 10.1016/j.gie.2007.12.046. PMID 18440381
- See also: research center of Sainte Justine Hospital — http://www.chu-sainte-justine.org/recherche/